CLINICAL TRIAL: NCT01950442
Title: Balloon Dilation of Malignant Strictures to Permit Complete Endoscopic Ultrasound Staging in Esophageal Cancer
Brief Title: Balloon Dilation to Permit Complete Endoscopic Ultrasound Staging in Esophageal Cancer
Acronym: CT0046
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CE13.118
Record Dates: First submitted 2013-09-23; First posted 2013-09-25 (Estimated); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Esophageal Cancer
Keywords: malignant strictures; esophageal staging
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Balloon dilation

SUMMARY:
Despite improvement in treatment-related morbidity and mortality, esophageal cancer is still one of the most lethal malignancies. Accurate staging is essential to establish prognosis and for patient management. Staging helps to determine if surgery, chemotherapy, radiation therapy, a combination of these, or a palliative approach is the most appropriate.

Endoscopic ultrasound techniques are becoming more and more popular. At Notre Dame Hospital, Centre Hospitalier de L'Universite de Montreal, all patients diagnosed with esophageal cancer undergo complete EUS staging. In selected patients, EUS is followed by EBUS during the same procedure, in order to examine all the lymph nodes near or far from the primary tumor amenable to EBUS guided trans-bronchial biopsy. In patients with a malignant esophageal stricture, we have preformed very gentle balloon dilation up to 14 mm. It is important to realize that this is not to achieve symptom resolution, but rather to allow the passage of the scope. We hypothesize that earlier reports of higher perforation rates were related to unnecessary aggressive dilation. Thus far, we have successfully dilated over 60 patients during the last four years (2009-2013) and were able to pass the scope and complete the examination in the vast majority of patients with no morbidity.

DETAILED DESCRIPTION:
The gold standard for evaluating the local extension of esophageal cancer is endoscopic ultrasound (EUS). The tumor extension into the esophageal wall (T stage) is best assessed using EUS. Suspicious lymph nodes in the mediastinum and in lymph node basins drained by the tumor (N stage) can be biopsied through the esophagus with fine needle aspiration (FNA) to obtain pathologic confirmation. Computed tomography (CT) and positron-emission tomography (PET) are used for the assessment of metastatic disease(M stage). In selected patients with liver lesions, EUS can be utilized to biopsy these and confirm metastatic disease. In the absence of metastatic disease, the local extent of the disease is an important factor in making the decision between surgery alone, neoadjuvant chemo-radiotherapy followed by surgery, surgery followed by chemoradiation or inoperability.

A difficult situation is encountered in patients with malignant strictures, where the EUS scope cannot be passed across the tumor and into the distal esophagus and stomach. There are several problems with this situation. The first is the inability to assess the complete T stage of the tumor. This can be associated with under T-staging. Also, the mediastinal and intra-abdominal lymph nodes distal to the tumor are not assessed, and this can also lead to inaccurate staging (N and M understaging). Patients with high grade malignant strictures have a worse prognosis, and therefore accurate staging and appropriate application of therapeutic options becomes paramount in providing the optimal treatment plan for this population.

To circumvent the problem of incomplete staging due to tight malignant strictures, one option that has been recently employed is gentle dilation of the malignant stricture, enough to allow passage of the scope. It is important to stress that the purpose is not to relieve any symptoms of dysphagia, but rather to allow passage of the scope to evaluate the TNM stage. There has been mixed results with regards to the safety of this technique. The following table summarizes the results of the studies evaluating dilation during endoscopic staging of esophageal cancer. The earliest reports quote a high complication rate of 24%, specifically related to perforation10. In the current era and with more experience gained in endoscopic diagnostic and therapeutic applications, there have been more reports of patients safely undergoing dilatation to permit complete endosonographic evaluation. The most recent studies report no perforations in their series. Except for the study performed by Pfau et al., the numbers are quite small with less than 40 patients in 3 of the studies. Furthermore, only one study by Wallace et al. reports any change in the staging offered by completing the EUS examination.

The study consists of a phase I clinical trial. All patients currently undergoing esophageal cancer staging in the Division of Thoracic Surgery at the CHUM will be approached for potential enrolment into the study. This staging is currently going on within the staging protocol for esophageal cancer and therefore is not a change in practise, however, patients refusing enrolment will not have there data included in the study database and their outcomes will not be used in any way for research protocols.

Patients with a malignant stricture that precludes passage of the dedicated endosonographic scope will comprise the study group. In this situation, an over-the-wire balloon dilation will be performed up to 14 mm. Patients in whom a standard adult gastroscope does not traverse the stricture, a pediatric gastrosocpe will be utilized in order to allow tumor traversal and guidewire placement into the stomach under endoscopic visualization. This will be performed in order to avoid dilating through the tumor and inadvertently causing a perforation. Once the dilation is complete, a complete EUS examination will be undertaken. EUS, followed by EBUS in selected patients with lymphadenopathy in the high mediastinal lymph nodes will be performed for staging.

All patients will undergo upright chest x-rays following their procedure in order to assess for pneumoperitoneum and pneumomediastinum. Patients will be discharged, as usual, following their procedure. Results will be discussed with them in a follow-up clinic appointment with their thoracic surgeon within 3 to 4 weeks of the procedure. Any procedure-related morbidity will be documented in the post-procedural period as well as at follow-up in the clinic. In patients sent from another hospital for EUS staging of esophageal cancer, which are not treated and followed at the CHUM, a 30 day telephone interview will be performed to assess for complications in the 30-day post-procedure period.

F. Data Points to be Collected

* Age
* Sex
* Comorbidties
* BMI
* Tumor location
* Tumor histology
* CT stage
* PET stage
* EUS T stage
* EUS N stage
* EUS M stage
* EUS lymph node FNA results
* EBUS lymph node FNA results
* Change in treatment plan based on completed EUS
* Procedural morbidity related to staging procedure
* 30-day morbidity related to staging procedure
* Pathologic staging, if available after undergoing surgical resection

Analysis will focus on:

1. Ability to complete an endosonographic examination after dilation
2. Safety profile of minimal dilation to allow passage of the EUS scopes
3. Change in treatment plan based on the completed endosonographic examination of esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven esophageal cancer
* Endoluminal esophageal mass without previous biopsy
* Medical suitability for endoscopic procedure
* Ability to consent

Exclusion Criteria:

* Patient on Coumadin (Warfarin), Plavix (Clopidogrel) or other anticoagulants with inability to stop medication for 5 days prior to procedure
* Tumors so tight that even a pediatric endoscope cannot traverse the stricture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2013-10; Primary Completion 2017-06 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Safety of gentle dilation | 10 months
  Examine the safety of gentle dilation of a malignant stricture to permit a complete endosonographic examination in patients with strictures not allowing passage of the EUS scope.
  Determine the proportion of patients that could undergo a complete EUS examination after dilation up to a maximum 14 mm.

SECONDARY OUTCOMES:
impact on staging | 10 months
  Examine the impact on staging gained by completing the EUS examination after dilation compared to the situation of non-dilation (incomplete staging due to non-passage of tumor).

CONTACTS AND LOCATIONS:
Overall Officials: Moishe Liberman, MD, PhD, Principal Investigator — CHUM-Centre Universitaire de Montreal
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Molina JC, Goudie E, Pollock C, Menezes V, Ferraro P, Lafontaine E, Martin J, Nasir B, Liberman M. Balloon Dilation for Endosonographic Staging in Esophageal Cancer: A Phase 1 Clinical Trial. Ann Thorac Surg. 2021 Apr;111(4):1150-1155. doi: 10.1016/j.athoracsur.2020.06.063. Epub 2020 Aug 29. PMID 32866480